CLINICAL TRIAL: NCT05012033
Title: Evaluation of High Dose Prednisolone Pharmacokinetics in the Acute and Chronic Setting
Acronym: EHD-Pred PK
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21HH6792
Record Dates: First submitted 2021-07-30; First posted 2021-08-19 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Thyroid Eye Disease; Vasculitis; COPD Exacerbation Acute; Asthma; Inflammatory Disease
MeSH Terms: conditions — Graves Ophthalmopathy; Vasculitis; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients started acutely on high dose prednisolone (>30mg for any inflammatory condition)
  Interventions: Other: No intervention - prednisolone is taken as part if routine clinical care.
- Group B: Patients on longer term anti-inflammatory doses of prednisolone to treat any medical condition warranting their use, including post COVID.
  Interventions: Other: No intervention - prednisolone is taken as part if routine clinical care.
- Group C: Patients receiving multiple high doses of methylprednisolone or dexamethasone in association with oral prednisolone.
  Interventions: Other: No intervention - prednisolone is taken as part if routine clinical care.

INTERVENTIONS:
Other: No intervention - prednisolone is taken as part if routine clinical care. — Prednisolone given orally prior to taking timed samples for levels

SUMMARY:
This is a pilot study to investigate serum prednisolone profiles in:

* Patients on high doses of prednisolone for any inflammatory disorder, both in the acute and chronic setting.
* Patients stepping up from or down to prednisolone therapy in association with a course of high dose methyl-prednisolone or dexamethasone.

The study will comprise 3 groups, including those started on high doses of prednisolone acutely in an inpatient or outpatient setting, participants on chronically high doses, and those receiving a several week course of high dose methylprednisolone or dexamethasone.

The study aims to measure prednisolone levels at a number of time points to investigate serum profile differences in those receiving prednisolone acutely compared with longer term steroid use. Further samples will be taken to characterise additional metabolic changes.

DETAILED DESCRIPTION:
Prednisolone is an anti-inflammatory drug widely used to reduce inflammation and immune activation in a number of medical conditions, including asthma, allergy, inflammatory and auto-immune conditions. Its therapeutic actions, however, are accompanied by several adverse side effects, which are more frequent following high doses and long term treatments. The aim is therefore to use the lowest effective dose or highest dose for the shortest treatment required.

It has been observed in a select number of patients on replacement prednisolone doses for adrenal insufficiency (AI) that serum prednisolone levels change over time, despite patients remaining on the same dose. It is currently unclear whether serum levels of prednisolone match the doses in patients taking high dose prednisolone, both in the acute and chronic setting, and whether the way in which prednisolone is metabolised is altered after receiving high doses for prolonged periods of time.

The rationale for the use of particular doses for particular conditions is not clear, and has been developed historically in the absence of individual patient data. It is possible that more tailored dosing of prednisolone will result in reduced side effects, and that the minimum possible dose may be weight related.

In addition, genetic and epigenetic factors may also play a role in the efficacy of prednisolone and in the risk of developing side effects, accounting for some of the inter-individual variation in drug response.

Further characterising this may help to create an evidence base to tailor anti-inflammatory doses and weaning regimens of synthetic glucocorticoids that avoid deleterious effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 75 years
* Male or female
* Participants who are otherwise healthy enough to participate, as determined by pre-study medical history
* Participants who are able and willing to give written informed consent to participate in the study
* Group A only: Patients requiring acute (<5 days) high dose (minimum 30mg) oral prednisolone therapy for antiinflammatory purposes in either an inpatient or outpatient setting.
* Group B only: Minimum of 1 month duration of high dose prednisolone (>30mg) if in the chronic use group.
* Group C only: Patients started on high dose methylprednisolone (>3 day course) or prolonged courses of dexamethasone.

Exclusion Criteria:

* Participants with a diagnosis of Type 1 or Type 2 diabetes mellitus.
* Unable to give informed consent.
* Taking supplements or herbal medications that the participant is unwilling or unable to stop prior to and during the study period e.g. St John's Wort (may decrease prednisolone levels), Cat's claw, Echinacea (immunomodulatory properties).
* Currently taking medications that alter CYP3A4 metabolism of glucocorticoids that the participant is unwilling or unable to stop prior to and during the study period e.g. phenytoin, phenobarbital, rifampicin, rifabutin, carbamazepine, primidone, aminogluethimide, itraconazole, ketoconazole, ciclosporin or ritonavir.
* Pregnancy. Females of child-bearing age will be asked to provide a urine sample for a pregnancy test at each visit.
* History of any medical, psychological or other condition, or use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study or compromise the safety of the participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving high dose prednisolone for any inflammatory disorder.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
To elucidate differences in prednisolone pharmacokinetics (in patients receiving high dose prednisolone acutely and in the chronic setting). | Pharmacokinetics measurements taken at the first and second visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  This will be assessed by determination of Cmax
To elucidate differences in prednisolone pharmacokinetics (in patients receiving high dose | Pharmacokinetics measurements taken at the first and second visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  This will be assessed by determination of Tmax
To elucidate differences in prednisolone pharmacokinetics (in patients receiving high dose | Pharmacokinetics measurements taken at the first and second visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  This will be assessed by determination of prednisolone half life and area under the curve values.
To elucidate differences in prednisolone pharmacokinetics (in patients receiving high dose | Pharmacokinetics measurements taken at the first and second visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  This will be assessed by determination of urinary steroid profiles.

SECONDARY OUTCOMES:
To elucidate further differences in metabolic profiles and glucocorticoid axis | Time points post prednisolone dose at 1st and 2nd visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  Assessed by review of bloods, including full blood count (FBC), renal profile, liver function tests (LFTs), creatine kinase (CK), Adrenocorticotropic hormone (ACTH), cortisol, cortisol binding globulin (CBG) and bicarbonate.
Exploratory Outcomes | Time points post prednisolone dose at 1st and 2nd visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  Metabolomic and metagenomic changes in plasma and urine to investigate inter-individual variation in prednisolone Immunology profiles - assessed by measurement and assessment of soluble immunological analytes and isolated white cell populations
  metabolism
Surrogate markers and risk factors for cardiovascular disease | On 1st and 2nd visits
  Anthropometric markers such as blood pressure
Surrogate markers and risk factors for cardiovascular disease | On 1st and 2nd visits
  Anthropometric markers such as heart rate
Surrogate markers and risk factors for cardiovascular disease | On 1st and 2nd visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  Anthropometric markers such as BMI
Surrogate markers and risk factors for cardiovascular disease | On 1st and 2nd visits. This will be of variable duration depending on duration of steroid treatment (5 days up to 2 years)
  Anthropometric markers such aswaist-hip circumference ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Meeran, MBBS BSc MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No